CLINICAL TRIAL: NCT06150547
Title: Pilot Imaging Study for CNS Metabolism
Brief Title: A Study of Metabolic Agents Following Brain Radiation
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 22-009871; NCI-2024-03176 (Other: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: CNS Malignancy
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Central Nervous System Malignant Tumor: Subjects may receive up to two CEST MRI's tests and/or up to two FDG PET. The physician will determine which test is appropriate based on your tumor type, past treatment history and research question. Tests will be completed at initial baseline visit and at least one other MRI/PET after the initial baseline, up to a maximum of four scans. Additionally, patients undergo finger-poke blood collection prior to receiving FDG on study.
  Interventions: Diagnostic Test: FDG Positron Emission Tomography; Diagnostic Test: Chemical Exchange Saturation Transfer Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: FDG Positron Emission Tomography — Imaging using an FDG radioactive tracer to look at the head.
  Other Names: FDG PET scan; fludeoxyglucose-18 (FDG) positron emission tomography (PET)
Diagnostic Test: Chemical Exchange Saturation Transfer Magnetic Resonance Imaging — A noninvasive diagnostic test for measuring biochemical changes in the brain, especially the presence of tumors.
  Other Names: CEST MRI

SUMMARY:
This study is being done to determine if CEST magnetic resonance imaging (MRI) and FDG PET are feasible techniques to detect metabolic differences between tumor and brain in patients with a brain tumor.

ELIGIBILITY:
Inclusion Criteria:

* Radiographic evidence or histopathologic confirmation of CNS malignancy, with or without prior resection.
* Provide written informed consent for the current study.
* Willing to undergo at least one MRI (and possibly more at PI discretion) with proton and/or phosphorus magnetic resonance spectroscopy analysis.

Exclusion Criteria:

* Vulnerable populations: pregnant or nursing women (Arm B exempt), prisoners, mentally handicapped.
* Cardiac pacemaker or artificial heart valve
* Metal plate, pin, or other metallic implant
* Intrauterine device, such as Copper-7 IUD
* Insulin or other drug pump
* Non-titanium aneurysm clips
* Previous gunshot wound
* Cochlear implant or other hearing device
* Employment history as a metalworker (had metal in eye)
* Permanent (tattoo) eye-liner
* For FDG-PET specifically: Fasting blood sugar level greater than 200mg/dl

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects identified as having a central nervous system malignant tumor undergoing routine care in the neuro-oncology practice at Mayo Clinic Rochester.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2023-12-27 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Number of subjects in whom glutamate metabolite is detected and measurable. | Baseline
  Number of subjects in whom glutamate metabolite is detected and measurable via CEST MRI in tumor, brain, and/or the ventricular space.
Number of subjects in whom n-acetylaspartate (NAA) metabolite is detected and measurable. | Baseline
  Number of subjects in whom n-acetylaspartate (NAA) metabolite is detected and measurable via CEST MRI in tumor, brain, and/or the ventricular space.

SECONDARY OUTCOMES:
Time required to perform the CEST MRI study and measure metabolites of interest | Duration of CEST MRI scan, approximately one to two hours.
  Total time expressed in minutes required to perform the CEST MRI study and measure metabolites of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Terry C Burns, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials